CLINICAL TRIAL: NCT06842264
Title: The Development and Validation of MRI-AI-based Predictive Models for csPCa
Status: Recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: prostatemodel19-29
Record Dates: First submitted 2025-02-11; First posted 2025-02-24 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer
Keywords: clinically-significant prostate cancer; artificial intelligence; magnetic resonance imaging; predictive model
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cohort 1: Cohort 1 comprises patients who underwent prostate magnetic resonance imaging (MRI) at Peking University First Hospital between January 2024 and December 2029, followed by an ultrasound-guided prostate biopsy.

SUMMARY:
This study retrospectively included patients who underwent prostate magnetic resonance imaging (MRI) and subsequent ultrasound-guided prostate biopsy at Peking University First Hospital from January 2019 to December 2023, and prospectively enrolls patients from January 2024 to December 2029. Clinical information such as age, PSA levels, PI-RADS scores, and digital rectal examination findings are collected. A well-performing artificial intelligence model is employed to measure prostate volume, transitional zone volume, and lesion volume using MRI images. Furthermore, prostate-specific antigen density (PSAD), transitional zone-based prostate-specific antigen density (TZ-PSAD) and lesion-based prostate-specific antigen density (lesion-PSAD) are calculated using prostate volume, transitional zone volume and lesion volume. Utilizing the aforementioned data, machine learning predictive models for clinically-significant prostate cancer (csPCa) are developed and validated.

DETAILED DESCRIPTION:
This study retrospectively included patients who underwent prostate magnetic resonance imaging (MRI) and subsequent ultrasound-guided prostate biopsy at Peking University First Hospital from January 2019 to December 2023, and prospectively enrolls patients from January 2024 to December 2029. Clinical information such as age, PSA levels, PI-RADS scores, and digital rectal examination findings are collected. A well-performing artificial intelligence model is employed to measure prostate volume, transitional zone volume, and lesion volume using MRI images. Furthermore, prostate-specific antigen density (PSAD), transitional zone-based prostate-specific antigen density (TZ-PSAD) and lesion-based prostate-specific antigen density (lesion-PSAD) are calculated using prostate volume, transitional zone volume and lesion volume. Utilizing the aforementioned data, machine learning predictive models for clinically-significant prostate cancer (csPCa) are developed and validated

ELIGIBILITY:
Inclusion Criteria:

* The interval between prostate MRI and biopsy within 3 months
* Integrity of related data

Exclusion Criteria:

* PSA less than 50ng/ml
* Any treatment for PCa prior to either MRI or biopsy, including radical prostatectomy, radiotherapy, chemotherapy, and endocrine therapy
* Previous history of surgical treatment or 5α-reductase inhibitor therapy for benign prostatic hyperplasia
* Subjects undergoing MRI with an indwelling urinary catheter or suprapubic catheter
* Inadequate quality of MRI images

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent prostate magnetic resonance imaging (MRI) at Peking University First Hospital between January 2024 and December 2029, followed by an ultrasound-guided prostate biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Biopsy pathology results | 1week after biopsy
  The pathology report will include the ISUP grade; if it is greater than or equal to 2, it is considered csPCa (clinically significant prostate cancer), otherwise, it is classified as non-csPCa.

CONTACTS AND LOCATIONS:
Overall Officials: Yi LIU, Principal Investigator — Dept. of Urology, Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, China